CLINICAL TRIAL: NCT06515119
Title: Efficacy of the Resources-Oriented Salutogenic (ROS) Intervention on Sense of Coherence Among Pre-diabetes Population: A Pilot Randomized Controlled Trial
Brief Title: Resources-Oriented Salutogenic (ROS) Intervention for Pre-diabetes
Acronym: ROS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSEARS20231206006
Record Dates: First submitted 2024-05-09; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-04

CONDITIONS: Sense of Coherence; Salutogenesis; PreDiabetes
Keywords: Salutogenesis; sense of coherence; resources; prediabetes
MeSH Terms: conditions — Prediabetic State | interventions — Methods

STUDY DESIGN:
Intervention Model Description: 66 prediabetes participants will be randomized into the intervention group and control group. Randomization will be conducted using the Research Randomizer Software and performed by a research team member who will not contact participants. Allocation will be concealed in sealed envelopes and revealed until trials commence, that is, after participants' submission of consent forms and completion of baseline assessments.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors who are uninvolved in other study phases will be unaware of group allocation. Participants will be advised not to disclose their group assignment to outcome assessors during the data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resources-oriented Salutogenic Intervention (Experimental): Intervention contents: Participants in the intervention group (IG) will receive online Resources-oriented Salutogenic intervention in the form of group lectures and in-session activity via Zoom meetings, and home activity via Facebook. Each group will have 7-8 participants. The intervention contents will provide information about resources and their utilization skills on health literacy related to prediabetes, healthy diet, exercise training, stress management, social support, and peer support. They will receive a) a resources booklet, b) "My Salutogenic Diary" for daily life recording, c) receive monthly telephone follow-ups.
  Intervention form: online group courses via Zoom meetings and Facebook. Intervention frequency and duration: 90 minutes per week, 8 weeks and two telephone follow-ups, once a month.
  Interventions: Behavioral: Resources-Oriented Salutogenic (ROS) intervention
- Usual Care (No Intervention): The control group (CG) will receive usual care (that is, general health education about lifestyle) on Facebook and undergo monthly educational follow-ups via Facebook messages to check the practical application of healthy lifestyle.

INTERVENTIONS:
Behavioral: Resources-Oriented Salutogenic (ROS) intervention — Participants in intervention group will receive an online ROS course via Zoom meeting, post daily salutogenic recordings and comments on Facebook. A closed Facebook group will be created to deliver resources booklet, zoom meeting links, as well as encourage participants share their daily salutogenic recording, give comments and thumps-up by group members.
  Arms: Resources-oriented Salutogenic Intervention

SUMMARY:
This pilot randomized control trial (RCT) is to assess whether the newly developed resources-oriented intervention is feasible and acceptable to people with pre-diabetes and has preliminary efficacy on sense of coherence (SoC).

The research questions are:

1. What are the key components (available resources and their utilization skills) of Resources-Oriented Salutogenic intervention in Chinese pre-diabetes population?
2. What are the feasibility and acceptability of ROS intervention among pre-diabetes population in China?
3. What is the preliminary efficacy of ROS intervention on improving sense of coherence, coping strategies, perceived stress, health literacy, and HbA1c on Chinese pre-diabetes population?

DETAILED DESCRIPTION:
Background:

General advice on lifestyle modification is given to people with pre-diabetes, but low participation and limitation of education time and location is noted in diabetes prevention programs and low SoC level still exists among pre-diabetes population. Salutogenesis-oriented interventions are effective on people with diabetes but none of such interventions have been designed and applied to people with pre-diabetes in China. People with pre-diabetes has not been educated to identify and utilize their available resources to cope with their stressful and unhealthy condition (pre-diabetes).

Objectives and methods: This study includes 3 phases:

Phase 1: ROS intervention components exploration for Chinese Pre-diabetes population Objectives: to explore preferred available resources for improving SoC among Chinese Pre-diabetes population.

Study design: A qualitative study. Individual in-depth semi-structured interviews guided by Salutogenic model will be conducted for approximately 40-60 min to explore the experience of coping with prediabetes, preferred General Resistance Resources (GRRs) and their utilizations after being diagnosed with prediabetes in Chinese pre-diabetes population.

Method: Purposive sampling will be used to select targeted population. The targeted population will be included: adults above 18 years, who have been diagnosed with pre-diabetes by medical staff or by undergoing HbA1c testing (5.7-6.4%). Sample size will be determined by the principle of data saturation, that is when no new relevant information or themes are observed in the data.

Phase 2: ROS intervention protocol development and refinement

Objectives:

1. to confirm the proposed key components of ROS intervention to be in line with professionals' expectations;
2. to refine the ROS intervention protocol

Study design: Content validity + qualitative study. Phase 2a: Six experts in diabetes prevention will be invited to assess the content validity of intervention protocol using a designed 10-item assessment form, aiming at achieving a satisfactory cut-off value of 0.83 in each item content validity index (i-CVI).

Phase 2b: The semi-structured interviews with focus group (4 participants in each group) aim to evaluate the readability, acceptability, and feasibility of the intervention protocol among prediabetes population in Hong Kong.

Method: For phase 2a, the inclusion criteria for experts will include: 1) have at least an expertise bachelor's degree; 2) have at least 3 years of working or research experience in their specialized area and be familiar with work in the field related to diabetes. Invitations will be extended via email, with a two-week response window for participation and form submission. For phase 2b, 12 prediabetes participants will be recruited from district health centers in Hong Kong. A doctoral student and a research assistant will conduct the 60-minute interview with participants via Zoom meeting to discuss words, sentences, or other specific contents with difficult to understand. All feedback from participants will help formulate the ROS intervention. The interview could be stopped until no new findings or information merged.

Phase 3: Preliminary assessment in Pilot RCT

Objectives:

1. to assess preliminary efficacy of ROS intervention on SoC, coping styles, perceived stress, health literacy, and HbA1c among prediabetes population in Hong Kong;
2. to explore their intervention experience.

Study design: a pilot RCT + a qualitative study nested within the pilot trial

Methods: For pilot RCT, 66 prediabetes participants will be randomized into the intervention group (IG) and control group (CG). Participants in IG will receive an online ROS course via Zoom meeting, post daily salutogenic recordings and comments on Facebook. While participants in CG will receive usual care (that is, general health education about lifestyle) in the Facebook and undergo monthly educational follow-ups via Facebook messages to check the practical application of healthy lifestyle. The primary outcome is SoC, and secondary outcomes include coping strategies, perceived stress, health literacy, and HbA1c, feasibility outcomes.

For a nested qualitative study, 10 participants with extreme SoC level (low and high) will be purposely selected to participate in the semi-structured interview. The SoC level will be assessed by SoC-13 scale depending on the score differences between baseline and post-intervention tests.

Data analysis:

For qualitative data, a six-step inductive thematic analysis will be used in Phase 1, while content analysis will be used in Phase 2 and a nested qualitative study in Phase 3.

For quantitative study, socio-demographic and feasibility data will be presented in absolute numbers and percentages for nominal (categorical) data, and Mean, and standard deviation for ratio (continuous) data or ordinal data. Homogeneity test for baseline will use Chi-square, Independent t-test, or Mann-Whitney U test. Generalized Estimating Equations will be used to analyze the efficacy differences in all primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria: Subjects are those with pre-diabetes and low or moderate level of sense of coherence.

1. prediabetes diagnosis: Pre-diabetes app score >= 8, considered as 'pre-diabetes' or 'at high-risk of diabetes'; then, HbA1c test result within 5.7% to 6.4% will be diagnosed as prediabetes.
2. low or moderate SoC level: SoC-13 scale score <= 74.
3. Chinese (Mandarin or Cantonese) or English and live in China,
4. could use Facebook and Zoom meeting app.

Exclusion Criteria:

Participants will be excluded if they:

1. have a history of diabetes, using hypoglycemic drugs, pregnancy, lactation, disability, or other physical limitations;
2. presence of serious health complications might affect the HbA1c level such as anemia, renal failure, liver disease;
3. participation in a similar intervention program within 3 months focusing on diabetes prevention in the past three months including educational workshops or courses, nutritional program, exercise program or mental health intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Sense of Coherence | Baseline; 8 weeks; 20 weeks
  SoC level of pre-diabetes population will be measured by 13-item Sense of Coherence Scale (SoC-13). It includes consists of 13 items in three domains: comprehensibility (item: 2,6,8,9,11), manageability (item: 3,5,10,13), and meaningfulness (item: 1,4,7,12). The 7-point Likert scale was used along with five reverse scoring items (item: 1,2,3,7,10). Higher scores indicate a higher level of SoC; a low level of SoC corresponded to SoC scores of 13-57, medium level referred to 58-74, and high SoC was 75-91.

SECONDARY OUTCOMES:
Diabetes risk | Baseline; 8 weeks; 20 weeks
  The pre-diabetes App is a convenient, non-invasive and straightforward tool for measuring diabetes risk. It includes the Chinese version of Finnish Diabetes Risk Score (FINDRISC) as well as the questions related to potential factors of diabetes like diabetes history, smoking, drinking, dietary pattern and physical activity engagement. The overall scores range from 0 to 26. The score of pre-diabetes app is greater than 8 in Chinese population indicating high-risk of diabetes.
Coping styles | Baseline; 8 weeks; 20 weeks
  The Simplified Copying Style Questionnaire (SCSQ) will be used to measure the pre-diabetes population's coping styles after diagnosed with high-risk of diabetes.This scale consisted of 20 items and two subscales: positive (12 items) and negative coping style (8 items), with a 4-point Likert scale from 0 (never) to 3 (frequently). Higher scores in subscales indicated that the respondents are to adopt positive or negative coping styles.
Perceived stress | Baseline; 8 weeks; 20 weeks
  The Perceived Stress Scale (PSS) will be used to measure the perception of stress in pre-diabetes population. The PSS-10 is a 10-item instrument with negative aspect (items 1,2,3,6,9,10) and positive aspect (items 4,5,7,8). This scale used a five-point Likert scale with scores ranging from 0 (never) to 4 (very often), with total scores from 0 to 20. Higher scores indicate higher perceived stress.
Diabetes literacy | Baseline; 8 weeks; 20 weeks
  The Chinese Health Literacy Scale for diabetes (CHLSD) will be used to measure the level of health literacy related to prediabetes. This scale consisted of 34 items and four sub-scales: remembering (18 items), understanding (7 items), applying (5 items) , analyzing (4 items). Two scores are given to the correct answer of each item. The CHLSD ranged from 0 to 68, with the total scores less than 48 indicating inadequate health literacy; the higher scores indicate the better health literacy. The Cronbach's alpha of four sub-scales in Chinese population is from 0.65 to 0.88.
Health promotion behaviors | Baseline; 8 weeks; 20 weeks
  The health promotion lifestyle profile-II (HPLP-II) will be used to measure health promotion behaviours of pre-diabetes population. A total of 52 items were measured using four-point Likert scale, with total score ranging from 52 to 208. The higher scores indicate better engagement in health-promoting behaviours. The total scores of low, moderate, high level correspond 52-104, 205-156, 157-208, respectively.
The glycated hemoglobin (HbA1c) test | Baseline; 20 weeks
  A portable HbAc1 test system by point-of-care testing (Cobas b101 system) will be used to measure HbAc1 levels.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Leung, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antonovsky, A. Health, stress, and coping: New perspectives on mental and physical well-being. San Francisco: 1979.
- [Background] Eriksson M. The Sense of Coherence: The Concept and Its Relationship to Health. 2022 Jan 1. In: Mittelmark MB, Bauer GF, Vaandrager L, Pelikan JM, Sagy S, Eriksson M, Lindstrom B, Meier Magistretti C, editors. The Handbook of Salutogenesis [Internet]. 2nd edition. Cham (CH): Springer; 2022. Chapter 9. Available from http://www.ncbi.nlm.nih.gov/books/NBK584067/ PMID 36121981
- [Background] Eriksson M, Lindstrom B. Validity of Antonovsky's sense of coherence scale: a systematic review. J Epidemiol Community Health. 2005 Jun;59(6):460-6. doi: 10.1136/jech.2003.018085. PMID 15911640
- [Background] Leung AY, Lou VW, Cheung MK, Chan SS, Chi I. Development and validation of Chinese Health Literacy Scale for Diabetes. J Clin Nurs. 2013 Aug;22(15-16):2090-9. doi: 10.1111/jocn.12018. Epub 2012 Nov 27. PMID 23186320
- [Background] Leung AY, Xu XY, Chau PH, Yu YTE, Cheung MK, Wong CK, Fong DY, Wong JY, Lam CL. A Mobile App for Identifying Individuals With Undiagnosed Diabetes and Prediabetes and for Promoting Behavior Change: 2-Year Prospective Study. JMIR Mhealth Uhealth. 2018 May 24;6(5):e10662. doi: 10.2196/10662. PMID 29793901
- [Background] Terry G, Hayfield N, Clarke V, et al. Thematic analysis. The SAGE handbook of qualitative research in psychology, 2017, 2(17-37): 25.
- [Background] Xie, Y. Reliability and validity of the simplified Coping Style Questionnaire. Chinese Journal of Clinical Psychology, 1998; 6(2), 114-115.
- [Background] Antonovsky A. Unraveling the mystery of health: How people manage stress and stay well. San Francisco. 1987;175.
- [Background] Leung DY, Lam TH, Chan SS. Three versions of Perceived Stress Scale: validation in a sample of Chinese cardiac patients who smoke. BMC Public Health. 2010 Aug 25;10:513. doi: 10.1186/1471-2458-10-513. PMID 20735860

DOCUMENTS (1):
  • Informed Consent Form (2024-03-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT06515119/ICF_000.pdf